CLINICAL TRIAL: NCT07241286
Title: Evaluation of the Effectiveness of Enhanced Recovery After Surgery (ERAS) Program in Pediatric Lung Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202504141RINE
Record Dates: First submitted 2025-10-02; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Lung Surgery; Enhanced Recovery After Surgery, ERAS; Pediatric
Keywords: Thoracoscopic; Partial resection; pediatric; infant; ERAS; VATS; lobectomy; segmentectomy
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enhanced Recovery After Surgery, ERAS: During the study period, all enrolled patients will be managed according to our institution's consensus ERAS checklist for pediatric lung surgery.
  Interventions: Other: Enhanced Recovery After Surgery, ERAS

INTERVENTIONS:
Other: Enhanced Recovery After Surgery, ERAS — During the study period, all enrolled patients will be managed according to our institution's consensus checklist for pediatric lung surgery ERAS care. This includes ERAS education, preoperative assessment, fasting guidance, prophylaxis for nausea and vomiting, standardized anesthesia and surgical protocols, preference for minimally invasive surgery, multimodal postoperative analgesia, and encouragement of early oral intake and mobilization.

SUMMARY:
This study aims to evaluate the clinical effectiveness of the Enhanced Recovery After Surgery (ERAS) program for pediatric lung surgery at our institution.

DETAILED DESCRIPTION:
Using a prospective cohort design, we will observe pediatric patients undergoing lung surgery following the implementation of the ERAS program as standard practice. Outcomes will be compared with a historical control group (2014-2023) to assess whether ERAS reduces hospital length of stay, lowers postoperative complication rates, accelerates recovery, and decreases healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent lung surgery at our hospital's Division of Pediatric Surgery

Exclusion Criteria:

* Patients who underwent multiple surgeries (including surgeries other than lung surgery) during the same hospitalization

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 0 to 18 years who underwent lung surgery at our institution. Eligible procedures were identified using treatment thoracoscopic lobectomy, thoracoscopic wedge or partial resection, and thoracoscopic segmentectomy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 30 days after surgery.
  Number of days from index operation to hospital discharge

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days after surgery.
  Incidence of postoperative complications, including prolonged air leak, pneumonia, surgical site infection, and other procedure-related events.
Duration of urinary catheter placement | From date of surgery to catheter removal (up to 30 days)
  Number of days with indwelling urinary catheter postoperatively.
Duration of chest tube drainage | From date of surgery to chest tube removal (up to 30 days).
  Number of days with thoracic drainage tube postoperatively.
Intensive care unit stay | From date of ICU admission to transfer out (up to 30 days).
  Number of days in ICU after surgery.
Postoperative pain | Daily assessment up to 7 days postoperatively.
  Pain intensity assessed by numeric rating scale (NRS)
Postoperative analgesic use | Daily assessment up to 7 days postoperatively.
  Total analgesic consumption.
30-day readmission or emergency department visit | Within 30 days post-discharge.
  Incidence of unplanned readmission or emergency department visit within 30 days after discharge.
Time to resumption of oral intake | From date of surgery to initiation of oral intake (up to 7 days).
  Interval from surgery to first tolerated oral feeding.
Hospital cost | From date of admission to discharge, up to 30 days
  Total hospitalization cost during the index admission.

OTHER OUTCOMES:
ERAS protocol adherence rate | Up to 30 days after surgery
  Proportion of ERAS protocol elements implemented per patient compared to total eligible elements.
Patient satisfaction with ERAS program | Up to 30 days after surgery.
  Satisfaction assessed by structured questionnaire at discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Children 2021, 8(12), 1154
- [Background] Ha D, Harris KT, Brockel MA, Rove KO. The role of enhanced recovery after surgery (ERAS) in promoting quality improvement and patient safety in pediatric urology. Front Urol. 2023 Sep 28;3:1275276. doi: 10.3389/fruro.2023.1275276. eCollection 2023. PMID 40778051